CLINICAL TRIAL: NCT02802904
Title: Multicountry Studies on the Effect of Positional Distribution of Fatty Acids at Triglyceride Backbone on Serum Lipids, Lipoprotein(a) and LDL-subclasses in Healthy Malaysian Volunteers
Acronym: MC1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malaysia Palm Oil Board (Other Government)
Collaborators: IMU University, Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: PD205/15- STUDY 1 (A)
Record Dates: First submitted 2016-06-02; First posted 2016-06-16 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Cardiovascular Risk Factor
Keywords: Healthy subjects

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Palm olein IV 64 (Experimental): Palm olein IV 64, n= 15, 4 weeks intervention
  Interventions: Other: Diet: Palm olein IV64
- Cocoa butter (Experimental): Cocoa butter, n= 15, 4 weeks intervention
  Interventions: Other: Diet: Cocoa butter
- Virgin olive oil (Experimental): Virgin olive oil, n= 15, 4 weeks intervention
  Interventions: Other: Diet: Virgin olive oil

INTERVENTIONS:
Other: Diet: Palm olein IV64 — Each subject received a palm olein-based run in diet for 2 weeks, followed by random assignment test fat Palm Olein IV64 which was incorporated into daily snacks (~50g of test fats, brownies (~15g test fat each) for breakfast and 4 pieces cookies (~5g test fat each) with low fat palm olein based background diet daily.
  Arms: Palm olein IV 64
Other: Diet: Cocoa butter — Each subject received a palm olein-based run in diet for 2 weeks, followed by random assignment test fat cocoa butter which was incorporated into daily snacks (~50g of test fats, brownies (~15g test fat each) for breakfast and 4 pieces cookies (~5g test fat each) with low fat palm olein based background diet daily.
  Arms: Cocoa butter
Other: Diet: Virgin olive oil — Each subject received a palm olein-based run in diet for 2 weeks, followed by random assignment test fat virgin olive oil which incorporated into daily snacks (~50g of test fats, brownies (~15g test fat each) for breakfast and 4 pieces cookies (~5g test fat each) with low fat palm olein based background diet daily.
  Arms: Virgin olive oil

SUMMARY:
Fats and oils are made up of >90% triacylglycerol fat molecules which consist of a glycerol backbone to which 3 esterified fatty acids are attached. The positions of fatty acid attachment are referred to by stereospecific numbers, sn -1, -2 and -3. There is existing evidence to show that vegetable oils having unsaturated fatty acids in the sn-2 position with predominantly palmitic acid (16:0) or stearic acid (18:0) in the sn-1 and sn-3 positions of fat molecules do not raise serum cholesterol levels. These observations have come to be known as or explained by the "sn-2 hypothesis". New evidence have also emerged to show that saturated fatty acids (16:0, 18:0) in the sn-1 and -3 positions reduces fat deposition in a rat model. In this proposed study, the effects on the outcome measures investigated of three test fats [namely palm olein IV64 (POP), virgin olive oil (OOO) and cocoa butter (POS)], with oleic acid primarily at the sn-2 position but differing amounts of palmitic, stearic and oleic acids at the sn-1/sn-3 positions of the triglyceride molecule, are investigated

DETAILED DESCRIPTION:
To investigate the effects of different dietary fats with primarily oleic acid in the sn-2 position on the cardiovascular risk profile in healthy Malaysian volunteers

ELIGIBILITY:
Inclusion criteria:

* Healthy adult male or female, aged 20-50 years
* BMI 18.5- 24.9 kg/m2 as per WHO Classification (1998)

Exclusion criteria:

* Hyperlipidemia (TC>6.2 mmol/L, TAG >2.0 mmol/L)
* History of chronic disease- type 2 DM, heart disease, cancer
* Habitual smokers (>2 sticks a day)
* Hypertensives: >140/90 mmHg
* On medication/nutraceuticals to reduce blood lipids, blood pressure
* Pregnant or lactating women
* Planned trip abroad/overseas during period of study

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Changes of Ratio of total cholesterol to HDL cholesterol (TC:HDL) | week 0 (baseline) and week 4
  analyzed enzymatically by Siemens Advia 2400 Chemistry Analyzer

SECONDARY OUTCOMES:
changes of serum HDL cholesterol | week 0 (baseline) and week 4
  analyzed enzymatically by Siemens Advia 2400 Chemistry Analyzer
changes of serum LDL cholesterol | week 0 (baseline) and week 4
  analyzed enzymatically by Siemens Advia 2400 Chemistry Analyzer
changes of serum Triacylglycerol (TAG) | week 0 (baseline) and week 4
  analyzed enzymatically by Siemens Advia 2400 Chemistry Analyzer
changes of serum non-esterified fatty acids (NEFA) | week 0 (baseline) and week 4
  analysed by ELISA kits
changes of serum LDL sub-fractions | week 0 (baseline) and week 4
  analysed with LIPOPRINT System
changes of serum Lp(a) | week 0 (baseline) and week 4
  analyzed enzymatically by Siemens Advia 2400 Chemistry Analyzer
changes of Blood pressure | week 0 (baseline) and week 4
  measured by blood pressure meter
Changes of body mass index (BMI) | week 0 (baseline) and week 4
  measured by Tanita Segmental Body Fat Analysis
changes of Waist circumference | week 0 (baseline) and week 4

CONTACTS AND LOCATIONS:
Overall Officials: Datuk Dr. Choo Yuen May, PhD, Study Chair — MPOB; Emeritus Prof. Datuk Dr. Augustine Ong Soon Hock, PhD, Study Chair — Malaysian Oil Scientists and Technologists' Association (MOSTA); Assoc Prof Dr Tony Ng Kock Wai, PhD, Principal Investigator — IMU; Dr Kanga Rani Selvaduray, PhD, Principal Investigator — MPOB; Radhika Loganathan, MSc, Principal Investigator — MPOB; Dr Darren Gouk Siew Wah, PhD, Principal Investigator — MPOB; Gowri Nagapan, MSc, Principal Investigator — MPOB

IPD SHARING:
Plan to Share IPD: Undecided